CLINICAL TRIAL: NCT06606470
Title: All Providers Better Communication Skills Program' (ABCs) Interprofessional Provider Education Randomized Controlled Trial
Brief Title: All Providers Better Communication Skills Program' (ABCs)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Health Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 17801
Record Dates: First submitted 2024-09-11; First posted 2024-09-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Education of Primary Care Clinicians; Palliative Care; Communication
Keywords: Palliative Care; Education; seriously ill communication; Observed Structured Clinical Examination (OSCE); Provider Training; Virtual learning
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: The study design is a prospective stepped wedge group - randomized controlled trial (SWGRT) of interprofessional health care providers (HCPs) who enroll in the ABCs program. In this trial design, half of the participants begin the study in the control condition as randomly assigned, and cross-over to the intervention condition at a pre-determined time points, so that both the intervention and control groups eventually receive the intervention. The primary comparison will be between the trial arms upon completion of a program by the initial intervention group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Full ABCs education program
  Interventions: Behavioral: All providers Better Communication Skills program' (ABCs) interprofessional provider education
- Control (No Intervention): No ABCs education program

INTERVENTIONS:
Behavioral: All providers Better Communication Skills program' (ABCs) interprofessional provider education — The 'All providers: Better Communication Skills program' (ABCs) is a virtual, person-centred education curriculum for interprofessional health care providers. The ABCs program adopts a blended format (i.e., participants engage in both asynchronous online modules [five] and synchronous interactive workshops [three]) that has relevance to learners and clinicians at all levels of training and practice. The ABCs program focuses on four essential elements of being a skillful communicator: principles of effective communication, conversation structure, communication skills, and reflective practice. The program consists of virtual modules that provide any clinician with practical tools, tips, and strategies to implement when communicating with seriously ill patients and their families. Terminology is clarified and consistent, the complexities of conversations are simplified and the fundamental approach and structure can be applied to different contexts.
  Arms: Intervention

SUMMARY:
High quality, person-centered communication for those living with serious illness benefits patients, families and clinicians. Evidence shows that clinicians rarely engage patients in these, sometimes challenging, discussions. Current education programs to build health care provider competency in serious illness communication are often inconsistent in defined purpose and use of terms. This education also tends to be oriented to treatments, not a person or do not cover the full range of difficult conversations between diagnosis and delivery of end-of-life care.

The ABCs program is an education intervention for health care providers that features a blended format of online modules and interactive virtual workshops, relevant to clinicians at all levels of training and practice. This study will examine the effectiveness of this training (over no training) for impacting provider competency and behavior change in serious illness communication. All participants in this study will receive the full ABCs training, but at different times. The overall intended impact of this program is to improve clinician confidence and satisfaction in having conversations with patients and families about serious illness. The ultimate goal of the ABCs program is to increase access to early palliative care by empowering more providers to initiate this care.

DETAILED DESCRIPTION:
Evidence shows that clinicians rarely engage patients in discussions about their serious illness and that there is a lack of training options to help health care providers develop these communication skills. By developing these skills, these conversations will be made easier, allowing patients to access a palliative approach to care earlier in their illness journey, providing them with the support and resources they need to manage their symptoms, alleviate their suffering, and improve their physical and mental health. This study will examine the ABCs education intervention that features a blended format of online modules and interactive virtual workshops, relevant to clinicians at all levels of training and practice, to build provider competency and comfort in serious illness communication.

The investigators developed the 'All providers: Better Communication Skills program' (ABCs), a virtual, person-centred education curriculum for interprofessional health care providers. This curriculum is a product of the collaboration among a large interdisciplinary team of palliative and end-of-life care clinicians, researchers, and educators, based on years of teaching advance care planning and goals of care discussions workshops with Hospice Palliative Care Ontario. The ABCs program adopts a blended format (i.e., participants engage in both asynchronous online modules [five] and synchronous interactive workshops [three]) that has relevance to learners and clinicians at all levels of training and practice. The investigators piloted this education program with medical learners and interdisciplinary health care providers with prior palliative care experience and still found that completion on the ABCs improved these participants self-reported confidence in initiating this communication and external rater assessments of their competency.

The ABCs program focuses on four essential elements of being a skillful communicator: principles of effective communication, conversation structure, communication skills, and reflective practice. The program consists of virtual modules that provide any clinician with practical tools, tips, and strategies to implement when communicating with seriously ill patients and their families. The ABCs program is intended to increase HCPs (particularly primary care providers) and medical learners' competency and comfort in having these, often difficult, conversations, while also encouraging them to initiate these discussions earlier in their patient's disease trajectory - moving a palliative approach to care further upstream. Terminology is clarified and consistent, the complexities of conversations are simplified and the fundamental approach and structure can be applied to different contexts.

The objective of this study is to complete a rigorous trial evaluating the impact of a communication skills curriculum for health care providers that addresses difficult conversations with seriously ill patients. The investigators aim to develop sustainable educational resources that can be administered virtually. Specially, the investigators will assess the impact of the ABCs education program on participant skill acquisition in communication and objective behavior change in simulated patient encounters. Secondly, the investigators will assess the impact of the education program on participant competency in communication from their own perspective and that of standardized patients with whom the participant has simulated encounters. The investigators will also measure participant satisfaction and perceived usefulness of the ABCs education program.

Potential participants across Canada will be informed about ABCs through advertising by the investigators partner stakeholders and organizations. The study design is a prospective stepped wedge group - randomized controlled trial (SWGRT) of interprofessional health care providers (HCPs) who enroll in the ABCs program. In this trial design, half of the participants begin the study in the control condition as randomly assigned, and cross-over to the intervention condition at a pre-determined time points, so that both the intervention and control groups eventually receive the intervention. The primary comparison will be between the trial arms upon completion of a program by the initial intervention group. This study will also measure the change among all participants from pre to post intervention.

ELIGIBILITY:
Inclusion Criteria:

All individuals that work in a health care provision capacity including health care professionals, care coordinators and administrators are eligible to enroll and participate in the ABCs study.

Exclusion Criteria:

Individuals, including patients, that do not work in a health care provision capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Clinical Encounter-Communications Tool (ACE-CT) | All groups: 1) From enrollment to start of Intervention Group ABCs education, 2) Post ABCs education for Intervention Group, at 4 months, 3) Post ABCs education for Control Group, at 8 months. Sample: 6 months post ABCs (14 months).
  The Assessment of Clinical Encounter-Communications Tool (ACE-CT) is completed by external raters of the recorded simulated practices, on a 5-point scale (1 to 5), with higher scores representing a better outcome. The ACE-CT is comprised of 14 items that were developed by the research team through a rigorous mixed methods Bayesian and Delphi process. This scale was derived from an extensive review of existing validated tools to measure quality of communication, including Communication in Oncology Questionnaire [Com-On], Family Meeting Communication Assessment Tool [FaMCAT] Comskil Coding System (CCS), Serious Illness Conversation Evaluation Exercise [SIC-Ex], and Gap-Kalamazoo Communication Skills Assessment Form. Item selection was based on the evidence of elements of HCP communication that are of high importance to patients and families and in which there are gaps in current experiences and practices.

SECONDARY OUTCOMES:
Self-Efficacy Questionnaire (SE-12) | All groups: 1) From enrollment to start of Intervention Group ABCs education, 2) Post ABCs education for Intervention Group, at 4 months, 3) Post ABCs education for Control Group, at 8 months. Sample: 6 months post ABCs (14 months).
  Completed by participants, the Self-Efficacy Questionnaire (SE-12) is a 12 item survey developed to measure the impact of communication skills training from the perspective of the participants. The SE-12 uses a 10-point scale (1 to 10), with higher scores representing a better outcome. This questionnaire has been validated and widely used in different settings, with different types of HCPs. The SE-12 has demonstrated internal consistency (Cronbach's α = 0.95) and response stability in test-retest reliability (Intraclass correlation agreement of 0.71). Scores were found to highly correlate with experience in clinical communication (P = 0.02).
End-of-life Professional Caregiver Survey (EPCS) | All groups: 1) From enrollment to start of Intervention Group ABCs education, 2) Post ABCs education for Intervention Group, at 4 months, 3) Post ABCs education for Control Group, at 8 months. Sample: 6 months post ABCs (14 months).
  Completed by participants, the End-of-life Professional Caregiver Survey (EPCS) is a 28-item scale developed to assess palliative care-specific educational needs related to three main subdomains: Effective Care Delivery (ECD 8-items); Patient and Family-Centered Communication (PFCC 12-items); and Cultural and Ethical Values (CEV 8-items). For the purposes of this study, the investigators will only include the Patient and Family-Centered Communication (PFCC) sub-domain. Each item is scored on a 5-point Likert scale ranging from 1 (lowest level of skill) to 5 (greatest level of skill), with higher scores representing a better outcome. Items represent care-provider comfort with a variety of situations related to palliative and EOL care. The EPCS covers all eight domains of the national palliative care guidelines and core lessons of physician-specific and nurse-specific end of life education curricula in the USA. The EPCS exhibits strong internal consistency (alpha = 0.96).
Blended Learning Usability Evaluation - Questionnaire (BLUE-Q) | Post ABCs education, at 4 months for Intervention Group, at 8 months for Control Group
  Completed by participants, the Blended Learning Usability Evaluation - Questionnaire (BLUE-Q) is a 31 item, three-part questionnaire that was developed and validated by members of this research team. The purpose of the BLUE-Q is to: evaluate the usability of blended learning programs, specifically those deployed across medical and health sciences education; systematize program evaluations for these interventions; and facilitate rigorous comparison between these different interventions. The BLUE-Q has a total of 23 Likert scale items (5-point scale, 1="Strongly Disagree" to 5="Strongly Agree", higher scores representing a better outcome) and 6 open-ended questions. The three parts of the BLUE-Q are: 1) pedagogical usability (i.e., the program content, learning objectives, and experience of learners with their instructors); 2) synchronous learning aspects; and 3) asynchronous learning aspects.
Qualitative Interviews | Post ABCs education, at 4 months for Intervention Group, at 8 months for Control Group
  In-depth interviews will be conducted via Zoom video communications application with select participants (15 to 25) in the ABCs, following completion of the intervention. This qualitative data collection will provide additional information on participant experience with the ABCs education program, applicability to practice, and learning context.
Questionnaire on Quality of Physician-Patient Interaction (QQPPI) | All groups: 1) From enrollment to start of Intervention Group ABCs education, 2) Post ABCs education for Intervention Group, at 4 months, 3) Post ABCs education for Control Group, at 8 months. Sample: 6 months post ABCs (14 months).
  Completed by Standardized Patients, the Questionnaire on Quality of Physician-Patient Interaction (QQPPI) is a 14 item, validated patient-facing rating scale of the for quality of physician communication. The QQPPI uses a 5-point scale (1 to 5), with higher scores representing a better outcome. This questionnaire is completed by patients to rate the quality of physician-patient interactions during outpatient care. The QQPPI demonstrates high internal consistency (Cronbach's α = 0.95) and significant correlations with other quality-related measures (Perceived Involvement in Care Scale [PICS] and Satisfaction with Decision Scale [SWD])
Feeling Heard and Understood scale | All groups: 1) From enrollment to start of Intervention Group ABCs education, 2) Post ABCs education for Intervention Group, at 4 months, 3) Post ABCs education for Control Group, at 8 months. Sample: 6 months post ABCs (14 months).
  Completed by Standardized Patients, the Feeling Heard and Understood scale is a 10 item, patient-reported quality measure for palliative care settings, on a 5-point scale (1 to 5) with higher scores representing a better outcome. The survey in intended for seriously ill patients to indicate the extent to which they feel feeling heard and understood by their care provider, have established trust in this individual, and that they perceive their care to have a whole-person orientation. The scale has been tested rigorously and found to exhibit validity and reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Hsien Seow, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Information deemed confidential.

REFERENCES:
- [Derived] Seow H, Arora AK, Bainbridge D, Jia Z, Steinberg L, Incardona N, Levine O, Sanders JJ, Simon J, des Ordons AR, Zhang K, Myers J. All providers Better Communication Skills (ABCs) program: protocol for a randomized controlled trial assessing communication training effectiveness with interprofessional clinicians. BMC Palliat Care. 2025 Nov 29;25(1):4. doi: 10.1186/s12904-025-01954-5. PMID 41318531